CLINICAL TRIAL: NCT04266821
Title: Establishing Clinical Utility of a New Diagnostic Test for Patients Suffering From Pain: A CPV® Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Ethos Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01ETH2020
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pain; Pain, Chronic
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study will enroll practicing primary care physicians in the US. Physicians are randomly assigned to either a control or intervention arm upon enrollment.
  All eligible and consented participants will complete two rounds of three patient simulations.
  The intervention arm only will receive educational material about the Ethos test in between these two rounds, and be provided simulated Ethos test results in the second round of simulated cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental-arm providers will complete two rounds of three simulated patient cases (CPVs) with two additions described in the next column:
  Interventions: Other: Experimental Arm
- Control (No Intervention): These providers will complete two rounds of three simulated patient cases (CPVs) only.

INTERVENTIONS:
Other: Experimental Arm — First, these providers will receive educational materials (e.g. a slide deck, mock test result and FAQ handout) meant to mimic what physicians will receive in the real-world market as they learn about the Ethos technology.
  Second, within each of their second-round cases, intervention-arm physicians only will receive simulated test results from the Ethos test at the clinically-appropriate point in each case.
  Arms: Experimental

SUMMARY:
This study will collect high-quality data on how practicing primary care physicians across the U.S. currently manage patients experiencing chronic pain and how the results of Ethos Laboratories' test change clinical decision making. To do so, this study leverages simulated patient cases called Clinical Performance and Value vignettes (CPVs) in a proven methodology to rapidly measure physician care decisions.

DETAILED DESCRIPTION:
This study will collect high-quality randomized controlled data from a nationally representative sample of practicing physicians, specifically primary care physicians and pain specialists, to determine how they currently manage patients with pain and how the results of Ethos' test change their clinical decision making. Data from this study will better illuminate the clinical use cases in which the Ethos test has the most significant impact on clinical decision making (and thus the largest clinical utility) and the physician characteristics (e.g., age, practice setting, training) associated with practice change.

The study is a prospective cohort trial with six steps:

1. Enrollment: The study will enroll an estimated 166 practicing primary care physicians who practice in the U.S. and are determined to be eligible by an eligibility screener.
2. Provider survey: Once providers are enrolled in the study, they will be asked to complete a questionnaire describing their practice and professional background.
3. Randomization: The 166 physicians will be randomized into equally-sized control and intervention arms.
4. CPVs (First Round): Physicians will complete three randomly-assigned CPV patient simulations. Cases will be identical across the intervention and control arms. All interactive cases are presented on an online platform, and are accessible via unique weblinks and any internet-connected computer.
5. Intervention education: Intervention-arm physicians will receive educational materials describing the clinical validation and use cases of the Ethos test. This material will replicate what physicians would receive as part of an actual marketing push introducing them to the Ethos test. These materials may be comprised of a slide deck, fact sheet, webinar, and/or case studies.
6. CPVs (Second Round): All participating physicians will then be asked to complete three additional CPV patient simulations. The cases are given to the doctors in a random order. Cases will be identical across the intervention and control arms, except that the intervention arm will receive Ethos test results at an appropriate point in each simulated case in the post-intervention round. Control arm physicians will continue to have access to standard of care diagnostic tools, but not the Ethos test results.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified physician for at least two years
2. Averaging at least 20 hours per week of clinical and patient care duties over the last six months
3. At least 15% of patient panel with chronic pain
4. Prescribes opioids
5. Practicing in the U.S.
6. English speaking
7. Access to the internet
8. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Practicing in an academic setting
3. Unable to access the internet
4. Not practicing in the U.S.
5. Not averaging at least 20 hours per week of clinical or patient care duties over the last six months
6. Less than 15% of panel with chronic pain
7. Does not prescribe opioids
8. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
CPV-measured pre-/post-difference in quality score between intervention and control physicians | 2-4 weeks
  Physicians completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the pre-/post-difference in these scores between control physicians using standard of care diagnostic tools and intervention physicians with access to Ethos test results, including by use case types
CPV-measured differences in evidence-based decisions made by intervention physicians and control physicians between rounds 1 and 2 | 2-4 weeks
  Physicians completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess differences in evidence-based decisions made by intervention physicians and control physicians between rounds 1 and 2, including by use case types
CPV-measured cost difference | 2-4 weeks
  Difference in cost of care between control and intervention physicians, including by use case types. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm on their CPVs, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs.)

SECONDARY OUTCOMES:
CPV-measured baseline variation | 1 week
  Physicians completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — President, QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgon TB, Cox-Chapman J, Czarnecki C, Kropp R, Guerriere R, Paculdo D, Peabody JW. Engaging Primary Care Providers to Reduce Unwanted Clinical Variation and Support ACO Cost and Quality Goals: A Unique Provider-Payer Collaboration. Popul Health Manag. 2019 Aug;22(4):321-329. doi: 10.1089/pop.2018.0111. Epub 2018 Oct 17. PMID 30328782
- [Background] Peabody J, Martin M, DeMaria L, Florentino J, Paculdo D, Paul M, Vanzo R, Wassman ER, Burgon T. Clinical Utility of a Comprehensive, Whole Genome CMA Testing Platform in Pediatrics: A Prospective Randomized Controlled Trial of Simulated Patients in Physician Practices. PLoS One. 2016 Dec 30;11(12):e0169064. doi: 10.1371/journal.pone.0169064. eCollection 2016. PMID 28036350
- [Background] Peabody JW, Strand V, Shimkhada R, Lee R, Chernoff D. Impact of rheumatoid arthritis disease activity test on clinical practice. PLoS One. 2013 May 7;8(5):e63215. doi: 10.1371/journal.pone.0063215. Print 2013. PMID 23667587
- [Background] Solon O, Woo K, Quimbo SA, Shimkhada R, Florentino J, Peabody JW. A novel method for measuring health care system performance: experience from QIDS in the Philippines. Health Policy Plan. 2009 May;24(3):167-74. doi: 10.1093/heapol/czp003. Epub 2009 Feb 18. PMID 19224955